CLINICAL TRIAL: NCT01257256
Title: Health Service Administration China Medical University
Brief Title: Investigating the Relationships Among Illness Cognition, Social Support, Stress, and Emotional Reactions of Infertile Patients
Acronym: HSA-246
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Jong-Yi Wang, China Medical University Hospital
Other Study IDs: CMU-DMR99-IRB-246
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Infertile Patients
Keywords: infertile patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- infertile patients: male infertile patients(ICD-9:606),female infertile patients(ICD-9:628)

SUMMARY:
The current study attempted to explore the relationships among stressors (cognitions of illness, socioeconomic status, social support, marital stressor, social stressor, etc), perceived stress level, and emotional reactions (anxiety and depression) of infertile patients and to propose the measurement and structural models of infertile aniexty and depression.

DETAILED DESCRIPTION:
The current study attempted to explore the relationships among stressors (cognitions of illness, socioeconomic status, social support, marital stressor, social stressor, etc), perceived stress level, and emotional reactions (anxiety and depression) of infertile patients and to propose the measurement and structural models of infertile aniexty and depression.

Structural Equation Modeling (SEM) will be utilized through AMOS 17 to analyze the data, construct the initial model, and afterward present the modified structural model of the psychological responses for infertile patients.

ELIGIBILITY:
Inclusion Criteria:male infertile patients(ICD-9:606) and female infertile patients(ICD-9:628).

Exclusion Criteria:non-infertile patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: simple random sampling
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan